CLINICAL TRIAL: NCT05018247
Title: A Prospective, Randomized Trial of Early Revascularization in Stable Ischemic Heart Disease Guided by Positron Emission Tomography of Artery Specific Integrated Comprehensive Quantitative Myocardial Perfusion
Brief Title: Early Revascularization in Stable Ischemic Heart Disease Using P.E.T. Imaging
Acronym: PETREVASC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated prematurely due to closure of the PET imaging facility
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, K.Lance Gould, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20211835
Record Dates: First submitted 2021-08-10; First posted 2021-08-24 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Heart Disease
Keywords: Positron Emission Tomography; PET scan
MeSH Terms: conditions — Myocardial Ischemia | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: After randomization, patients will receive urgent revascularization combined with Optimal Medical Treatment or Optimal Medical Treatment with delayed revascularization. Following the initial PET scan, randomization and treatment, each group will undergo a second PET scan at the 3-4 month mark and a third PET scan at the one year mark. At their first follow-up visit (3-4 month mark), patients in the OMT with delayed revascularization group will be offered the option of continued medical treatment or elective revascularization consistent with informed patient preference and clinical judgement. Patients, in consultation with their physicians, may elect to undergo revascularization at any time thereafter.
Masking Description: Study personnel and subjects will not be blinded. All core lab measurements, comparisons, and statistical analysis will be blinded to group assignment by blinded coding of PET images. Two volunteers who are not involved in the study in any way to create randomization envelopes with each arm. The study staff volunteers for randomization assignment will:
  Create a randomization list with two arms (52 per arm). Create 104 sequential envelopes which will contain a paper with the assignment based on the randomization list.
  The sequential randomization envelopes will be kept in the site PI's locked office thereby allowing for randomization immediately after consent is obtained. The randomization arm will be shared with the research team and the subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urgent revascularization with Optimal Medical Therapy (Active Comparator): Revascularization will be performed via either Percutaneous Coronary Intervention or Coronary Artery Bypass Graft, and the selection of the specific procedure will be at the discretion of the patient and their physician(s). Patients will be followed for one year after randomization. Follow-up visits will occur at Baseline, Day 105, and Day 365. At each visit, a rest-stress PET assessment will be performed, and adverse events related to study procedures and cardiac disease will be captured.
  Interventions: Procedure: Revascularization by Coronary Artery Bypass Graft or Percutaneous Coronary Intervention
- Optimal Medical Treatment with delayed revascularization (Other): OMT without revascularization for a minimum of approximately 105 days if clinically stable. At their first follow-up visit (Day 105±20), patients will be offered the option of continued medical treatment or elective revascularization consistent with informed patient preference and clinical judgement. Patients, in consultation with their physicians, may elect to undergo revascularization at any time thereafter and will be followed for one year after randomization. Follow-up visits will occur at Baseline, Day 105, and Day 365. At each visit, a rest-stress PET assessment will be performed, and adverse events related to study procedures and cardiac disease will be captured.
  Interventions: Procedure: Revascularization by Coronary Artery Bypass Graft or Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Revascularization by Coronary Artery Bypass Graft or Percutaneous Coronary Intervention — Urgent revascularization via CABG or PCI combined with Optimal Medical Treatment

SUMMARY:
To compare the impact of revascularization and Optimal Medical Treatment (OMT) on the extent of severely reduced coronary flow capacity in stable ischemic heart disease.

DETAILED DESCRIPTION:
The initial Positron Emission Tomography (PET) scan will be performed as part of clinical practice. If the patient is a potential candidate for the study, the patient will be screened for inclusion and exclusion criteria. After being informed about the study potential risks, all patients giving written informed consent will be randomized into one of two groups: Urgent revascularization combined with Optimal Medical Treatment (OMT) or OMT with delayed revascularization. Following the initial PET scan, randomization and treatment, each group will undergo a second PET scan at the 3-4 month mark and a third PET scan at the one year mark. Some crossover may occur with the two groups. The OMT without urgent revascularization patients will remain in that group, if clinically stable, up to three months. At their first follow-up visit (Day 105±20), patients will be offered the option of continued medical treatment or elective revascularization consistent with informed patient preference and clinical judgement. Patients, in consultation with their physicians, may elect to undergo revascularization at any time thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Stable ischemic heart disease as determined by an investigator.
3. Areas of severely reduced CFC or relative stress images on the Rentrop diagnostic PET MPI consistent with clinical judgement as follows:

   • PETs with a defect on rest relative images of ≤60% of max for ≤5% of LV (no large scar) plus: i. ≥2% of LV with CFCblue* or ii. ≥10% of LV with CFCgreen* plus at least one pixel with CFCblue*

   *CFCblue is defined as a dipyridamole induced stress flow ≤ 0.83 ml/min/g of myocardium and a CFR ≤ 1.27. CFCgreen is defined as a dipyridamole induced stress flow ≤1.09 and >0.83 ml/min/g of myocardium and a CFR ≤1.60 and >1.27.
4. Willing to comply with the follow-up schedule of the trial.
5. Subject must sign the informed consent in English or Spanish.

Exclusion Criteria:

1. Any conditions that may compromise or prevent the necessary imaging requirements.
2. Less than one-year life expectancy.
3. Currently pregnant or planning to become pregnant during the course of the study.
4. Any other issues that the Investigator believes may interfere with treatment or follow-up.
5. Subjects who lack capacity to consent for themselves.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the % of left ventricle (LV) with Coronary Flow Capacity (CFC)blue. | Baseline and Day 105+20
  CFCblue is defined as a dipyridamole induced stress flow ≤ 0.83 ml/min/g of myocardium and a CFR ≤ 1.27.
Change from baseline in the % of left ventricle (LV) with Coronary Flow Capacity (CFC)green. | Baseline and Day 105+20
  CFCgreen is defined as a dipyridamole induced stress flow ≤1.09 and >0.83 ml/min/g of myocardium and a CFR ≤1.60 and >1.27.

SECONDARY OUTCOMES:
Change in % of LV with CFCblue. | Baseline and Day 105 +20 and Day 365+30
  Change in % in Left Ventricle with Coronary Flow Capacity blue.
Change in % of LV with CFCgreen. | Baseline and Day 105 +20 and Day 365+30
  Change in % of Left Ventricle with Coronary Flow Capacity green.
Change in CFC histogram distribution. | Baseline and Day 105 +20 and Day 365+30
  Change in Coronary Flow Capacity histogram distribution.
Change in minimum quadrant average CFR. | Baseline and Day 105 +20 and Day 365+30
  Change in minimum quadrant average Coronary Flow Reserve.
Change in minimum quadrant average stress ml/min/g. | Baseline and Day 105 +20 and Day 365+30
  Minimum quadrant average stress changes during PET.
Change in minimum stress relative quadrant average. | Baseline and Day 105 +20 and Day 365+30
  Change in relative minimum uptake on stress images.
Change in global CFR. | Baseline and Day 105 +20 and Day 365+30
  Change in global Coronary Flow Reserve.
Change in specific iso-contour defect size & its average CFR. | Baseline and Day 105 +20 and Day 365+30
  Change in specific iso-contour defect size & its average Coronary Flow Reserve.
Change in DEFECT stress ml/min/g. | Baseline and Day 105 +20 and Day 365+30
  Change of absolute flow in ml/min/g in the defect during stress.
Change in DEFECT relative stress. | Baseline and Day 105 +20 and Day 365+30
  Change in size and severity of stress induced perfusion defects during stress.
Changes in an additional 120 PET flow fields. | Baseline and Day 105 +20 and Day 365+30
  Changes in 120 PET flow fields derived in the CORE lab comparing Rentrop PETs with reprocessed PETs at University of Texas Health Science Center Houston
Rate of adverse events | Baseline and Day 105 +20 and Day 365+30
  Rate of major adverse cardiovascular events (defined as death from cardiovascular causes, myocardial infarction, or hospitalization for unstable angina, heart failure, or resuscitated cardiac arrest).
Rate of safety events. | Baseline and Day 105 +20 and Day 365+30
  Rate of safety events during the course of the trial such as death or adverse effects.
Rate of procedure-related adverse events | Baseline and Day 105 +20 and Day 365+30
  Rate of procedure-related adverse events such as death from cardiovascular causes, myocardial infarction, or hospitalization for unstable angina, heart failure, or resuscitated cardiac arrest.

CONTACTS AND LOCATIONS:
Overall Officials: K. Lance Gould, MD, Principal Investigator — UT Health Science Center Houston
Locations (1):
- Gramercy Cardiac Diagnostic Services, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No